CLINICAL TRIAL: NCT05564390
Title: Master Screening and Reassessment Protocol (MSRP) for the NCI MyeloMATCH Clinical Trials
Brief Title: MYELOMATCH: A Screening Study to Assign People With Myeloid Cancer to a Treatment Study or Standard of Care Treatment Within myeloMATCH (MyeloMATCH Screening Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NCI-2022-07006; NCI-2022-07006 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MYELOMATCH (Other: SWOG); MYELOMATCH (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic/Myeloproliferative Neoplasm; Acute Myeloid Leukemia Post Cytotoxic Therapy; Acute Myeloid Leukemia, Myelodysplasia-Related; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myeloproliferative Disorders; Myelodysplastic Syndromes | interventions — Stem Cell Transplantation; Azacitidine; Practice Guidelines as Topic; Standard of Care; Biopsy; Specimen Handling; Busulfan; X-Rays; Cytarabine; Daunorubicin; decitabine and cedazuridine drug combination; enasidenib; fludarabine; Gemtuzumab; gilteritinib; CPX-351; Injections; Liposomes; Melphalan; olutasidenib; Magnetic Resonance Spectroscopy; Whole-Body Irradiation; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (34):
- MM1MDS-A01 Regimen 1 (ASTX727) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR, CRL, or CRh at the end of cycle 6 may cross-over to Regimen 2. Patients who experience CR, PR, or SD any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to TAP. Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine
- MM1MDS-A01 Regimen 2 (ASTX727, enasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5 and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience CR, PR, or SD any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to TAP. Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Enasidenib
- MM1OA-EA02 Regimen 1 (azacitidine, venetoclax) (Experimental): INDUCTION: Patients receive azacitidine IV or SC on days 1-7 of each cycle and venetoclax PO on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy and aspiration as well as blood sample collection on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Venetoclax
- MM1OA-EA02 Regimen 2 (azacitidine, venetoclax, gilteritinib) (Experimental): INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax and gilteritinib PO on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-7 and gilteritinib PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy and aspiration as well as blood sample collection on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Gilteritinib; Drug: Venetoclax
- MM1OA-EA02 Regimen 3 (azacitidine, venetoclax, gilteritinib) (Experimental): INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28, and gilteritinib PO on days 8-21 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-14 and gilteritinib PO on days 8-21 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo bone marrow biopsy and aspiration as well as blood sample collection on the trial.
  Interventions: Drug: Azacitidine; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Gilteritinib; Drug: Venetoclax
- MM1OA-MDS-A05 Cohort A, Arm 1 (ASTX727, venetoclax) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 of each cycle and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- MM1OA-MDS-A05 Cohort A,Arm 2 (ASTX727,venetoclax,olutasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5 of each cycle, venetoclax PO QD on days 1-28 of each cycle, and olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Olutasidenib; Drug: Venetoclax
- MM1OA-MDS-A05 Cohort B, Arm 3 (ASTX727, olutasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5 of each cycle and olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Olutasidenib
- MM1OA-MDS-A05 Cohort B, Arm 4 (ASTX727) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients without CR after cycle 6 may then cross-over to Arm 3. Patients with CR, as well as patients without CR but deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine
- MM1OA-MDS-A05 Cohort C (olutasidenib) (Experimental): Patients receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Olutasidenib
- MM1OA-S03 Arm 1 (ASTX727, venetoclax) (Active Comparator): Patients receive ASTX727 PO QD on days 1-5 and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow aspiration, and bone marrow biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Venetoclax
- MM1OA-S03 Arm 2 (ASTX727, venetoclax, enasidenib) (Experimental): Patients receive ASTX727 PO QD on days 1-5, venetoclax PO QD on days 1-28, and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow aspiration, and bone marrow biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Decitabine and Cedazuridine; Drug: Enasidenib; Drug: Venetoclax
- MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy) (Active Comparator): Patients receive gemtuzumab ozogamicin IV on days 1 and 4, cytarabine IV, continuously, on days 1-7 and daunorubicin IV on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or MUGA scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Gemtuzumab Ozogamicin; Procedure: Multigated Acquisition Scan
- MM1YA-A04 Regimen 2 (venetoclax, chemotherapy) (Experimental): Patients receive gemtuzumab ozogamicin IV on days 1 and 4, cytarabine IV, continuously, on days 1-7 and daunorubicin IV on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or MUGA scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- MM1YA-CTG01 Arm I (daunorubicin, cytarabine, venetoclax) (Experimental): Patients receive daunorubicin IV on days 2-4, cytarabine IV continuously on days 2-8, and venetoclax PO QD on days 1-11. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of daunorubicin IV on days 2-3, cytarabine IV continuously on days 2-6, and venetoclax PO QD on days 1-8. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Venetoclax
- MM1YA-CTG01 Arm II (azacitidine, venetoclax) (Experimental): Patients receive azacitidine IV or SC on days 1-7 or days 1-5 and 8-9 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for a total of 2 cycles, in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Venetoclax
- MM1YA-CTG01 Arm III (daunorubicin, cytarabine) (Active Comparator): Patients receive daunorubicin IV on days 1-3 and cytarabine IV, continuously, on days 1-7. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of cytarabine IV, continuously, on days 1-5 and daunorubicin IV on days 1-2. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride
- MM1YA-S01 Arm I (cytarabine, daunorubicin) (Active Comparator): Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV on days 1-3 per standard approach of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 1-5 and daunorubicin IV on days 1-2. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax) (Experimental): Patients receive cytarabine IV continuously on days 2-8 and daunorubicin IV on days 2-4 with venetoclax PO on days 1-11 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 2-6 and daunorubicin IV on days 2-3 with venetoclax PO on days 1-8. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- MM1YA-S01 Arm III (azacitidine, venetoclax) (Experimental): Patients receive azacitidine SC or IV on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- MM1YA-S01 Arm IV (Vyxeos) (Experimental): Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Echocardiography Test; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Multigated Acquisition Scan
- MM1YA-S01 Arm V (Vyxeos, venetoclax) (Experimental): Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 and venetoclax PO on days 1-14 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3 and venetoclax PO on days 1-7. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Echocardiography Test; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- MM2YA-EA01 Arm A (cytarabine) (Active Comparator): Patients receive cytarabine IV on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Drug: Cytarabine; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- MM2YA-EA01 Arm B (cytarabine, venetoclax) (Experimental): Patients receive cytarabine IV and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Drug: Cytarabine; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- MM2YA-EA01 Arm C (Vyxeos, venetoclax) (Experimental): Patients receive Vyxeos IV and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Procedure: Biopsy Procedure; Procedure: Echocardiography Test; Drug: Liposome-encapsulated Daunorubicin-Cytarabine; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- MM2YA-EA01 Arm D (azacitidine, venetoclax) (Experimental): Patients receive azacitidine IV or SC and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.
  Interventions: Drug: Azacitidine; Procedure: Biopsy Procedure; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax
- MM3TCT-A03 Conditioning 1A (matched donors with venetoclax) (Experimental): Patients receive venetoclax PO QD on days -10 to -2, fludarabine IV on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or BID on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Busulfan; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Venetoclax
- MM3TCT-A03 Conditioning 1B (matched donors with placebo) (Placebo Comparator): Patients receive placebo PO QD on days -10 to -2, fludarabine IV on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or BID on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Drug: Busulfan; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Drug: Placebo Administration; Procedure: Positron Emission Tomography
- MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax) (Experimental): Patients receive venetoclax PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Radiation: Total-Body Irradiation; Drug: Venetoclax
- MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo) (Placebo Comparator): Patients receive placebo PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Melphalan; Drug: Placebo Administration; Procedure: Positron Emission Tomography; Radiation: Total-Body Irradiation
- MM3TCT-A03 Maintenance I (venetoclax) (Experimental): Patients receive venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Multigated Acquisition Scan; Procedure: Positron Emission Tomography; Drug: Venetoclax
- MM3TCT-A03 Maintenance II (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo PET scan and/or CT scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Placebo Administration; Procedure: Positron Emission Tomography
- Screening (mutation carrier screening) (Experimental): Patients undergo bone marrow aspiration and collection of blood on study. Patients' bone marrow and blood specimens undergo rapid genetic testing. Patients are then assigned to a specific substudy containing a therapy targeted to the patient's mutational profile. If there is no targetable mutation, the patient is placed on a substudy testing novel combinations that do not contain a target-specific drug. Patients who are not eligible for any MYELOMATCH substudy are assigned to TAP.
  Interventions: Procedure: Mutation Carrier Screening
- TAP (SOC treatment, mutation carrier screening) (Experimental): Patients continue SOC treatment and undergo continued bone marrow aspiration and blood collection for possible future substudy assignment.
  Interventions: Other: Best Practice; Procedure: Mutation Carrier Screening

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Given IV
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
  Arms: MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo)
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: MM1OA-EA02 Regimen 1 (azacitidine, venetoclax); MM1OA-EA02 Regimen 2 (azacitidine, venetoclax, gilteritinib); MM1OA-EA02 Regimen 3 (azacitidine, venetoclax, gilteritinib); MM1YA-CTG01 Arm II (azacitidine, venetoclax); MM1YA-S01 Arm III (azacitidine, venetoclax); MM2YA-EA01 Arm D (azacitidine, venetoclax)
Other: Best Practice — Receive SOC treatment
  Other Names: standard of care; standard therapy
  Arms: MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); TAP (SOC treatment, mutation carrier screening)
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
  Arms: MM1OA-EA02 Regimen 1 (azacitidine, venetoclax); MM1OA-EA02 Regimen 2 (azacitidine, venetoclax, gilteritinib); MM1OA-EA02 Regimen 3 (azacitidine, venetoclax, gilteritinib); MM2YA-EA01 Arm A (cytarabine); MM2YA-EA01 Arm B (cytarabine, venetoclax); MM2YA-EA01 Arm C (Vyxeos, venetoclax); MM2YA-EA01 Arm D (azacitidine, venetoclax)
Procedure: Biospecimen Collection — Undergo collection of blood, urine, and/or buccal swab samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: MM1MDS-A01 Regimen 1 (ASTX727); MM1MDS-A01 Regimen 2 (ASTX727, enasidenib); MM1OA-EA02 Regimen 1 (azacitidine, venetoclax); MM1OA-EA02 Regimen 2 (azacitidine, venetoclax, gilteritinib); MM1OA-EA02 Regimen 3 (azacitidine, venetoclax, gilteritinib); MM1OA-MDS-A05 Cohort A, Arm 1 (ASTX727, venetoclax); MM1OA-MDS-A05 Cohort A,Arm 2 (ASTX727,venetoclax,olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 3 (ASTX727, olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 4 (ASTX727); MM1OA-MDS-A05 Cohort C (olutasidenib); MM1OA-S03 Arm 1 (ASTX727, venetoclax); MM1OA-S03 Arm 2 (ASTX727, venetoclax, enasidenib); MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM1YA-CTG01 Arm I (daunorubicin, cytarabine, venetoclax); MM1YA-CTG01 Arm II (azacitidine, venetoclax); MM1YA-CTG01 Arm III (daunorubicin, cytarabine); MM1YA-S01 Arm I (cytarabine, daunorubicin); MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax); MM1YA-S01 Arm III (azacitidine, venetoclax); MM1YA-S01 Arm IV (Vyxeos); MM1YA-S01 Arm V (Vyxeos, venetoclax); MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo); MM3TCT-A03 Maintenance I (venetoclax); MM3TCT-A03 Maintenance II (placebo)
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
  Arms: MM1MDS-A01 Regimen 1 (ASTX727); MM1MDS-A01 Regimen 2 (ASTX727, enasidenib); MM1OA-MDS-A05 Cohort A, Arm 1 (ASTX727, venetoclax); MM1OA-MDS-A05 Cohort A,Arm 2 (ASTX727,venetoclax,olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 3 (ASTX727, olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 4 (ASTX727); MM1OA-MDS-A05 Cohort C (olutasidenib); MM1OA-S03 Arm 1 (ASTX727, venetoclax); MM1OA-S03 Arm 2 (ASTX727, venetoclax, enasidenib); MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM1YA-CTG01 Arm I (daunorubicin, cytarabine, venetoclax); MM1YA-CTG01 Arm II (azacitidine, venetoclax); MM1YA-CTG01 Arm III (daunorubicin, cytarabine); MM1YA-S01 Arm I (cytarabine, daunorubicin); MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax); MM1YA-S01 Arm III (azacitidine, venetoclax); MM1YA-S01 Arm IV (Vyxeos); MM1YA-S01 Arm V (Vyxeos, venetoclax)
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
  Arms: MM1MDS-A01 Regimen 1 (ASTX727); MM1MDS-A01 Regimen 2 (ASTX727, enasidenib); MM1OA-MDS-A05 Cohort A, Arm 1 (ASTX727, venetoclax); MM1OA-MDS-A05 Cohort A,Arm 2 (ASTX727,venetoclax,olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 3 (ASTX727, olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 4 (ASTX727); MM1OA-MDS-A05 Cohort C (olutasidenib); MM1OA-S03 Arm 1 (ASTX727, venetoclax); MM1OA-S03 Arm 2 (ASTX727, venetoclax, enasidenib); MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo); MM3TCT-A03 Maintenance I (venetoclax); MM3TCT-A03 Maintenance II (placebo)
Drug: Busulfan — Given IV
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
  Arms: MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo)
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
  Arms: MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
  Arms: MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo); MM3TCT-A03 Maintenance I (venetoclax); MM3TCT-A03 Maintenance II (placebo)
Drug: Cytarabine — Given
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM1YA-CTG01 Arm I (daunorubicin, cytarabine, venetoclax); MM1YA-CTG01 Arm III (daunorubicin, cytarabine); MM1YA-S01 Arm I (cytarabine, daunorubicin); MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax); MM2YA-EA01 Arm A (cytarabine); MM2YA-EA01 Arm B (cytarabine, venetoclax)
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM1YA-CTG01 Arm I (daunorubicin, cytarabine, venetoclax); MM1YA-CTG01 Arm III (daunorubicin, cytarabine); MM1YA-S01 Arm I (cytarabine, daunorubicin); MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax)
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX 727; ASTX-727; ASTX727; C-DEC; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; DEC-C; Inaqovi; Inqovi
  Arms: MM1MDS-A01 Regimen 1 (ASTX727); MM1MDS-A01 Regimen 2 (ASTX727, enasidenib); MM1OA-MDS-A05 Cohort A, Arm 1 (ASTX727, venetoclax); MM1OA-MDS-A05 Cohort A,Arm 2 (ASTX727,venetoclax,olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 3 (ASTX727, olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 4 (ASTX727); MM1OA-S03 Arm 1 (ASTX727, venetoclax); MM1OA-S03 Arm 2 (ASTX727, venetoclax, enasidenib)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
  Arms: MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM1YA-S01 Arm I (cytarabine, daunorubicin); MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax); MM1YA-S01 Arm III (azacitidine, venetoclax); MM1YA-S01 Arm IV (Vyxeos); MM1YA-S01 Arm V (Vyxeos, venetoclax); MM2YA-EA01 Arm A (cytarabine); MM2YA-EA01 Arm B (cytarabine, venetoclax); MM2YA-EA01 Arm C (Vyxeos, venetoclax); MM2YA-EA01 Arm D (azacitidine, venetoclax); MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo)
Drug: Enasidenib — Given PO
  Other Names: AG 221; AG-221; AG221; CC-90007 Free Base
  Arms: MM1MDS-A01 Regimen 2 (ASTX727, enasidenib); MM1OA-S03 Arm 2 (ASTX727, venetoclax, enasidenib)
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
  Arms: MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo)
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
  Arms: MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy)
Drug: Gilteritinib — Given PO
  Other Names: ASP 2215; ASP-2215; ASP2215
  Arms: MM1OA-EA02 Regimen 2 (azacitidine, venetoclax, gilteritinib); MM1OA-EA02 Regimen 3 (azacitidine, venetoclax, gilteritinib)
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX 351; CPX-351; CPX351; Cytarabine and Daunorubicin Liposomal; Cytarabine-Daunorubicin Liposome for Injection; Daunorubicin and Cytarabine (Liposomal); Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos
  Arms: MM1YA-S01 Arm IV (Vyxeos); MM1YA-S01 Arm V (Vyxeos, venetoclax); MM2YA-EA01 Arm C (Vyxeos, venetoclax)
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
  Arms: MM1YA-A04 Regimen 1 (gemtuzumab ozogamicin, chemotherapy); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM1YA-S01 Arm I (cytarabine, daunorubicin); MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax); MM1YA-S01 Arm III (azacitidine, venetoclax); MM1YA-S01 Arm IV (Vyxeos); MM1YA-S01 Arm V (Vyxeos, venetoclax); MM2YA-EA01 Arm A (cytarabine); MM2YA-EA01 Arm B (cytarabine, venetoclax); MM2YA-EA01 Arm C (Vyxeos, venetoclax); MM2YA-EA01 Arm D (azacitidine, venetoclax); MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Maintenance I (venetoclax)
Procedure: Mutation Carrier Screening — Undergo rapid genetic testing
  Arms: Screening (mutation carrier screening); TAP (SOC treatment, mutation carrier screening)
Drug: Olutasidenib — Given PO
  Other Names: FT 2102; FT-2102; FT2102; IDH1-R132 Inhibitor FT-2102; Rezlidhia
  Arms: MM1OA-MDS-A05 Cohort A,Arm 2 (ASTX727,venetoclax,olutasidenib); MM1OA-MDS-A05 Cohort B, Arm 3 (ASTX727, olutasidenib); MM1OA-MDS-A05 Cohort C (olutasidenib)
Drug: Placebo Administration — Given PO
  Arms: MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo); MM3TCT-A03 Maintenance II (placebo)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
  Arms: MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 1B (matched donors with placebo); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo); MM3TCT-A03 Maintenance I (venetoclax); MM3TCT-A03 Maintenance II (placebo)
Radiation: Total-Body Irradiation — Undergo total body irradiation
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation
  Arms: MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Conditioning 2B (haplo/mismatch with placebo)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: MM1OA-EA02 Regimen 1 (azacitidine, venetoclax); MM1OA-EA02 Regimen 2 (azacitidine, venetoclax, gilteritinib); MM1OA-EA02 Regimen 3 (azacitidine, venetoclax, gilteritinib); MM1OA-MDS-A05 Cohort A, Arm 1 (ASTX727, venetoclax); MM1OA-MDS-A05 Cohort A,Arm 2 (ASTX727,venetoclax,olutasidenib); MM1OA-S03 Arm 1 (ASTX727, venetoclax); MM1OA-S03 Arm 2 (ASTX727, venetoclax, enasidenib); MM1YA-A04 Regimen 2 (venetoclax, chemotherapy); MM1YA-CTG01 Arm I (daunorubicin, cytarabine, venetoclax); MM1YA-CTG01 Arm II (azacitidine, venetoclax); MM1YA-S01 Arm II (cytarabine, daunorubicin, venetoclax); MM1YA-S01 Arm III (azacitidine, venetoclax); MM1YA-S01 Arm V (Vyxeos, venetoclax); MM2YA-EA01 Arm B (cytarabine, venetoclax); MM2YA-EA01 Arm C (Vyxeos, venetoclax); MM2YA-EA01 Arm D (azacitidine, venetoclax); MM3TCT-A03 Conditioning 1A (matched donors with venetoclax); MM3TCT-A03 Conditioning 2A (haplo/mismatch with venetoclax); MM3TCT-A03 Maintenance I (venetoclax)

SUMMARY:
This MyeloMATCH Master Screening and Reassessment Protocol (MSRP) evaluates the use of a screening tool and specific laboratory tests to help improve participants' ability to register to clinical trials throughout the course of their myeloid cancer (acute myeloid leukemia or myelodysplastic syndrome) treatment. This study involves testing patients' bone marrow and blood for certain biomarkers. A biomarker (sometimes called a marker) is any molecule in the body that can be measured. Doctors look at markers to learn what is happening in the body. Knowing about certain markers can give doctors more information about what is driving the cancer and how to treat it. Testing patients' bone marrow and blood will show doctors if patients have markers that specific drugs can target. The marker testing in this study will let doctors know if they can match patients with a treatment study (myeloMATCH clinical trial) that tests treatment for the type of cancer they have or continue standard of care treatment with their doctor on the Tier Advancement Pathway (TAP).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Screening and Reassessment (MSRP): To evaluate the feasibility of MATCHBox receiving and organizing all data needed for assignment to a myeloMATCH clinical trial or Tier Advancement Pathway (TAP) within 72 hours of MDNet receipt of all required specimens for initial therapy and within 10 days for subsequent therapy.

II. Tier Advancement Pathway (TAP): To enable participants who are not matched to an investigational myeloMATCH treatment substudy to receive standard of care (SOC) while remaining on the MSRP to maintain access to later tiers of treatment substudies.

SECONDARY OBJECTIVES:

I. Screening and Reassessment (MSRP):

Ia. To describe the time to generation of all data required for treatment substudy (or TAP) assignment, time to treatment substudy (or TAP) assignment, percent assigned to a myeloMATCH treatment substudy, and the percent of screened participants who register to a myeloMATCH investigational treatment substudy or are assigned to TAP:

Iai. Separately within each tier of myeloMATCH treatment substudy and analogous TAP assignment; Ibi. Separately within each clinical basket of myeloMATCH treatment substudies; Ici. Over time, across and within the categories above.

II. Tier Advancement Pathway (TAP):

IIa. To evaluate participants for assignment to higher tier treatment substudies within myeloMATCH; IIb. To describe, within tier- and basket- levels of TAP, measurable residual disease (MRD) rates and clonal evolution; IIc. To describe, within tier- and basket- levels of TAP, remission status and overall survival of participants who receive standard of care therapy; IId. To obtain MDNet specimens for translational medicine and biobanking.

OUTLINE:

REGISTRATION: Patients undergo bone marrow aspiration and collection of blood on study. Patients' bone marrow and blood specimens undergo rapid genetic testing. Patients are then assigned to a specific substudy containing a therapy targeted to the patient's mutational profile. If there is no targetable mutation, the patient is placed on a substudy testing novel combinations that do not contain a target-specific drug. Patients who are not eligible for any MYELOMATCH substudy are assigned to TAP.

TAP: Patients continue SOC treatment and undergo continued bone marrow aspiration and blood collection for possible future substudy assignment.

TREATMENT: Patients are assigned to a specific treatment substudy.

MM1YA-CTG01: Younger patients (age 18-59 years) with intermediate risk acute myeloid leukemia (AML) are randomized to 1 of 3 arms.

ARM I: Patients receive daunorubicin intravenously (IV) on days 2-4, cytarabine IV continuously on days 2-8, and venetoclax orally (PO) once per day (QD) on days 1-11. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of daunorubicin IV on days 2-3, cytarabine IV continuously on days 2-6, and venetoclax PO QD on days 1-8. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.

ARM II: Patients receive azacitidine IV or subcutaneously (SC) on days 1-7 or days 1-5 and 8-9 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for a total of 2 cycles, in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.

ARM III: Patients receive daunorubicin IV on days 1-3 and cytarabine IV, continuously, on days 1-7. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of cytarabine IV, continuously, on days 1-5 and daunorubicin IV on days 1-2. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.

MM1YA-S01: Younger patients (age 18-59 years) with high-risk AML are randomized to 1 of 5 arms.

ARM I: Patients receive cytarabine IV continuously on days 1-7 and daunorubicin IV on days 1-3 per standard approach of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 1-5 and daunorubicin IV on days 1-2. Patients undergo echocardiography (ECHO) or multigated acquisition (MUGA) scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM II: Patients receive cytarabine IV continuously on days 2-8 and daunorubicin IV on days 2-4 with venetoclax PO on days 1-11 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of cytarabine IV continuously on days 2-6 and daunorubicin IV on days 2-3 with venetoclax PO on days 1-8. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM III: Patients receive azacitidine SC or IV on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM IV: Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

ARM V: Patients receive daunorubicin and cytarabine liposome IV over 90 minutes on days 1, 3, and 5 and venetoclax PO on days 1-14 of each cycle. Cycles repeat every 28 days for 1 cycle in the absence of disease progression or unacceptable toxicity. Patients may receive an additional cycle of daunorubicin and cytarabine liposome IV over 90 minutes on days 1 and 3 and venetoclax PO on days 1-7. Patients undergo ECHO or MUGA scan during screening. Patients also undergo a bone marrow aspiration and collection of blood throughout the trial.

MM2YA-EA01: Younger patients (age 18-59 years) with AML or secondary AML who have completed a tier 1 MyeloMATCH treatment study with complete remission (CR) or CR with partial hematologic recovery (CRh) and have detectable minimal residual disease (MRD) (> 0.1%) are randomized to 1 of 4 arms.

ARM A: Patients receive cytarabine IV on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.

ARM B: Patients receive cytarabine IV and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.

ARM C: Patients receive Vyxeos IV and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.

ARM D: Patients receive azacitidine IV or SC and venetoclax PO on study. Patients undergo bone marrow aspiration and biopsy on study. Patients may also undergo ECHO and/or MUGA as clinically indicated.

MM1OA-EA02: Patients are randomized to 1 of 3 regimens.

REGIMEN 1:

INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

REGIMEN 2:

INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax and gilteritinib PO on days 1-28 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-7 and gilteritinib PO on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

REGIMEN 3:

INDUCTION: Patients receive azacitidine IV or SC on days 1-7 and venetoclax PO on days 1-28, and gilteritinib PO on days 8-21 of each cycle. Treatment repeats every 28 days for up to 2 cycles or until patient achieves remission, whichever comes first, in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive azacitidine IV or SC on days 1-5, venetoclax PO on days 1-14 and gilteritinib PO on days 8-21 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

MM1MDS-A01: Patients are randomized to 1 of 2 regimens.

REGIMEN 1: Patients receive ASTX727 PO once daily (QD) on days 1-5 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who do not achieve a CR, CRL, or CRh at the end of cycle 6 may cross-over to Regimen 1. Patients who experience CR, PR, or stable disease (SD) any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to TAP. Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.

REGIMEN 2: Patients receive ASTX727 PO QD on days 1-5 and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience CR, PR, or SD any time after 4 cycles of treatment may be reassessed in order to go to a higher myeloMATCH tier assignment or to TAP. Patients also undergo bone marrow biopsy and aspiration throughout the study. Patients may also undergo optional buccal swab on study, and/or optional additional bone marrow aspiration and blood sample collection on study and at disease progression.

MM1OA-S03: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive ASTX727 PO QD on days 1-5 and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow aspiration, and bone marrow biopsy throughout the trial.

ARM 2: Patients receive ASTX727 PO QD on days 1-5, venetoclax PO QD on days 1-28, and enasidenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, bone marrow aspiration, and bone marrow biopsy throughout the trial.

MM1YA-A04: Patients are randomized to 1 of 2 regimens.

REGIMEN 1: Patients receive gemtuzumab ozogamicin IV on days 1 and 4, cytarabine IV, continuously, on days 1-7 and daunorubicin IV on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or MUGA scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.

REGIMEN 2: Patients receive venetoclax PO QD on days 1-11, cytarabine IV, continuously, on days 2-8 and daunorubicin IV on days 2-4 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or MUGA scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.

MM3TCT-A03: Patients with matched donors are randomized to conditioning 1A or 1B. Patients with haploidentical or mismatched unrelated donors are randomized to conditioning 2A or 2B.

CONDITIONING 1A: Patients receive venetoclax PO QD on days -10 to -2, fludarabine IV on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or twice daily (BID) on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

CONDITIONING 1B: Patients receive placebo PO QD on days -10 to -2, fludarabine IV on days -6 or -5 to -2 and busulfan IV on days -3 to -2 or BID on days -5 to -2 or melphalan IV on day -2. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

CONDITIONING 2A: Patients receive venetoclax PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

CONDITIONING 2B: Patients receive placebo PO QD on days -10 to -2, melphalan IV on day -6, fludarabine IV on days -5 to -2 and undergo total body irradiation once on day -1. Patients then receive hematopoietic cell transplant IV on day 0. Treatment is given in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: All patients without evidence of relapse at day +100 are re-randomized to maintenance I or II.

MAINTENANCE I: Patients receive venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE II: Patients receive placebo PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 1 year post transplant (9 cycles) in the absence of disease progression or unacceptable toxicity.

Patients undergo chest x-ray, echocardiography or MUGA during screening, and bone marrow biopsy and blood, urine and buccal swab collection throughout the study. Patients may also undergo positron emission tomography (PET) scan and/or computed tomography (CT) scan throughout the study.

MM1OA-MDS-A05: Patients are assigned to 1 of 3 cohorts.

COHORT A: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive ASTX727 PO QD on days 1-5 of each cycle and venetoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

ARM 2: Patients receive ASTX727 PO QD on days 1-5 of each cycle, venetoclax PO QD on days 1-28 of each cycle, and olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR, CRh, or CRi after cycle 4 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

COHORT B: Patients are randomized to 1 of 2 arms.

ARM 3: Patients receive ASTX727 PO QD on days 1-5 of each cycle and olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with CR continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

ARM 4: Patients receive ASTX727 PO QD on days 1-5 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients without CR after cycle 6 may then cross-over to Arm 3. Patients with CR, as well as patients without CR but deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

COHORT C: Patients receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients deriving clinical benefit after cycle 6 continue treatment cycles every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy/aspiration and collection of blood samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be suspected to have previously untreated acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS). Participants with AML cannot have a history of previously treated myeloproliferative neoplasms (MPN) or MDS.
* Participants must be >= 18 years of age.
* Participants must not have received prior anti-cancer therapy for AML or MDS.

  * Note: Hydroxyurea to control the white blood cell count (WBC) is allowed.
  * Note: Prior erythroid stimulating agent (ESA) is not considered prior therapy for the purposes of eligibility. Participants must not be currently receiving any cytarabine-containing therapy other than up to 1 g/m^2 of cytarabine, which is allowed for urgent cytoreduction.
* Participants are allowed prior use of hydroxyurea, all-trans retinoic acid (ATRA), BCR-ABL directed tyrosine kinase inhibitor, erythropoiesis-stimulating agent, thrombopoietin receptor agonist and lenalidomide, with a maximum limit of 1 month of exposure.

  * Note: Participants receiving hydroxyurea prior to treatment substudy or TAP assignment must agree to discontinue hydroxyurea within 24 hours before beginning substudy or TAP treatment.
* Participants must not have a prior or concurrent malignancy that requires concurrent anti-cancer therapy

  * Note: active hormonal therapy is allowed
* Participants must have a Zubrod Performance Status evaluation within 28 days prior to registration.
* Participants must agree to have translational medicine specimens submitted.
* Participants must be offered the opportunity to participate in specimen banking.

  * Note: Specimens must be collected and submitted following the initial paper-based process and subsequently via the Precision Medicine Specimen Tracking Forms in Medidata Rave instance for the MyeloMATCH MSRP.
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines.

  * Note: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.
* The master screening and reassessment protocol (MSRP) should only be used in sites where the relevant AML treatment substudies are open or if the site is willing to follow the MSRP Tier Advancement Pathway (TAP) for patients in the event that the site does not have the relevant study open and transfer to another site that does have the study open. For example, if a site does not have a myeloMATCH Tier 1 study for older AML open for enrollment, such older AML patients should only be consented for the MSRP if the site is willing to treat the patient with standard of care on TAP or is willing to transfer the patient to a center with a study open that the patient would otherwise match to.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2029-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Timing of treatment Substudy or Tier Advancement Pathway (TAP) assignment | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will evaluate the feasibility of MATCHBox generating all data needed for assignment to a myeloMATCH clinical trial or determination that no assignment is available, within 72 hours of MDNet receipt of specimens for initial therapy and within 10 days for subsequent therapy. For first treatment assignment and separately for each subsequent treatment assignments: every 50 participants for the first 250 participants and then every 100 participants thereafter, the proportion of participants (cumulative and new participants since prior analysis) with all MDNet data needed to determine a treatment assignment within 72 hours for first assignment and 10 days for subsequent assignments after the MDNet receives specimens will be tallied.

SECONDARY OUTCOMES:
Time to MDNet generating all data required for treatment substudy or TAP assignment | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will be assessed within each tier of clinical trials, within each clinical basket of clinical trials, and over time (since last report and in 6 month intervals from study opening).
Time to treatment substudy or TAP assignment | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will be assessed within each tier of clinical trials, within each clinical basket of clinical trials, and over time (since last report and in 6 month intervals from study opening).
Percent assigned to a myeloMATCH clinical trial | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will be assessed within each tier of clinical trials, within each clinical basket of clinical trials, and over time (since last report and in 6 month intervals from study opening).
Percent of screened participants who register to a treatment substudy | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will be assessed within each tier of clinical trials, within each clinical basket of clinical trials, and over time (since last report and in 6 month intervals from study opening).
Assignment to higher tier treatment substudies within myeloMATCH | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will be assessed within each tier of clinical trials, within each clinical basket of clinical trials, and over time (since last report and in 6 month intervals from study opening).
Adverse events | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will be assessed within each tier of clinical trials, within each clinical basket of clinical trials, and over time (since last report and in 6 month intervals from study opening).
Minimal residual disease (MRD) response | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  MRD response is based on flow cytometry studies performed by the MDnet.
Time-to-event outcomes for exploratory analysis | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Will be assessed within each tier of clinical trials, within each clinical basket of clinical trials, and over time (since last report and in 6 month intervals from study opening).
Performance status | Within 72 hours of MDNet receipt of specimens for initial therapy or within 10 days for subsequent therapy
  Participants will be graded according to the Zubrod performance status scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jerald P Radich, Principal Investigator — SWOG Cancer Research Network
Locations (327):
- United States (315):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Yale University, New Haven, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Healthcare Mission Cancer and Blood - Pella, Pella, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - MaineHealth Cancer Care and IV Therapy - Brunswick, Brunswick, Maine
  - Mid Coast Hospital, Brunswick, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (10):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Tiong IS, Loo S. Targeting Measurable Residual Disease (MRD) in Acute Myeloid Leukemia (AML): Moving beyond Prognostication. Int J Mol Sci. 2023 Mar 1;24(5):4790. doi: 10.3390/ijms24054790. PMID 36902217